CLINICAL TRIAL: NCT02404168
Title: Evaluation of Repeatability of Lamotrigine Pharmacokinetics in Epileptic Patients
Brief Title: BEEP Follow Up: Evaluation of Repeatability of Lamotrigine Pharmacokinetics in Epileptic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, James E Polli, Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HP-00063848
Record Dates: First submitted 2015-03-17; First posted 2015-03-31 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- lamotrigine brand tablet1 (Active Comparator): lamotrigine tablet Lamictal
  Interventions: Drug: lamotrigine (brand Lamictal)
- lamotrigine generic tablet1 (Experimental): lamotrigine tablet Teva
  Interventions: Drug: lamotrigine (generic Teva)
- lamotrigine brand tablet2 (Active Comparator): lamotrigine tablet Lamictal
  Interventions: Drug: lamotrigine (brand Lamictal)
- lamotrigine generic tablet2 (Experimental): lamotrigine tablet Teva
  Interventions: Drug: lamotrigine (generic Teva)

INTERVENTIONS:
Drug: lamotrigine (brand Lamictal) — an anti-epileptic drug (brand)
  Other Names: Lamictal
  Arms: lamotrigine brand tablet1; lamotrigine brand tablet2
Drug: lamotrigine (generic Teva) — an anti-epileptic drug (brand)
  Other Names: generic lamotrigine
  Arms: lamotrigine generic tablet1; lamotrigine generic tablet2

SUMMARY:
The prior BEEP study involved patients being switched between brand and generic in a very structured manner. Other secondary comparisons were also made (i.e. any differences in adverse effects and seizure control). Some subjects were more disparate than other, in terms of generic being similar to brand. In this follow up study, BEEP subjects that showed disparate results will be tested again to assess reproducibility of disparate results.

DETAILED DESCRIPTION:
This is an double-blind, multiple-dose, full replicate design, pharmacokinetic study of lamotrigine in "enriched" patients with epilepsy who previously participated in HP-00048923. LAMICTAL 100mg tablets and the most commonly used generic lamotrigine 100mg tablet (from Teva) will be compared pharmacokinetically.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent and was enrolled in previous BEEP study.
* Subject is male or female between 18 and 76 years of age inclusive.
* Subject has a diagnosis of epilepsy with simple partial seizures and/or complex partial seizures, with or without secondary generalization or primary generalized seizures
* Subject has been maintained on a stable dose regimen of anti-epileptic drugs (AEDs), including lamotrigine at 200mg, 400mg, or 600mg total daily dosage divided BID for at least 8 weeks prior to Visit 1 and during the screening period
* Subject is willing to be switched between brand and generic lamotrigine
* Subject is an acceptable candidate for venipuncture
* Subject is willing to stop all OTC medications for 24 hours prior to and during 12 hour study visits

Exclusion Criteria:

* Subject is currently participating or has participated within the last 2 months in any trial of an investigational drug or experimental device
* Subject has a history of status epilepticus within the 12 month period prior to Visit 1.
* Subject has any medical condition, which in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in the trial
* Subject has any psychiatric condition, which in the opinion of the investigator, could jeopardize the subject's health or would compromise the subject's ability to participate in this trial or confound the interpretation of the trial data
* Subject has known hypersensitivity to lamotrigine
* Subject has a medical condition that impacts drug absorption (e.g. gastric bypass surgery), including routine use (i.e.

daily or weekly) use of acid blockers, antacids, anti-diarrhea, stimulants, appetite suppressants, or anti nausea medication or other drugs that modulate GI function

* Subject has any history of alcohol or drug abuse within the previous two years
* Subject has acute or subacutely progressive CNS disease
* Subject has moderate or severe liver impairment as assessed by alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels ≥5 times the upper limit of normal (ULN).
* Subject has moderate or severe renal impairment as assessed by creatinine clearance lower than 50mL/min, using the Cockcroft-Gault formula
* Female subjects of childbearing potential will not be eligible to participate who are unwilling or unable to use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: condom with spermicide, diaphragm with spermicide, IUD without progesterone, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence
* Female subject is pregnant or nursing
* Female subject is using hormonal contraceptive precautions including progesterone-coated IUD
* Subjects is using hormonal replacement therapy
* Subject is unwilling or unable to maintain their approximate daily smoking use during the study
* Subject is using rifampin or other non-AED that strongly modulates lamotrigine levels
* addition to lamotrigine and/or vagus nerve stimulation and/or intermittent benzodiazepine use (e.g. lorazepam, diazepam, clonazepam), subject is taking more than two concomitant AEDs
* Subject is not willing or able to be adherent to study protocol (e.g. dosing of lamotrigine and any interacting comedication).

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2016-01-18 (Actual); Study Completion 2016-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Background] Andermann F, Duh MS, Gosselin A, Paradis PE. Compulsory generic switching of antiepileptic drugs: high switchback rates to branded compounds compared with other drug classes. Epilepsia. 2007 Mar;48(3):464-9. doi: 10.1111/j.1528-1167.2007.01007.x. PMID 17346246

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine Tablet: Sequence: generic first, then brand, then brand, and then generic. Each of the four arms will be about two weeks in duration. During the study, subjects will receive their on-going therapeutic lamotrigine regimen of either 200mg, 400mg, or 600mg total daily dosage, divided in twice-a-day doses (i.e. every 12 hours). In the study, 100mg lamotrigine tablets (brand or generic) will be dispensed to the subject at the start of each study arm.
Period: Overall Study
Arm/Group | Lamotrigine Tablet
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Lamotrigine Tablet: Sequence: generic first, then brand, then brand, and then generic
Arm/Group | Lamotrigine Tablet
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 48 [22 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: pharmacokinetic exposure (ng*hr/ml). Pharmacokinetic (PK) blood levels will be drawn at the schedule times: immediately prior to lamotrigine administration, then after drug administration at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, and 12.0 hr.
Time Frame: 0-12hr
Measure: Mean (Standard Error); unit: ng*hr/ml
Groups:
- Active Comparator: Lamotrigine Brand: lamotrigine tablet Lamictal
- Experimental: Lamotrigine Generic: lamotrigine tablet Teva
Arm/Group | Active Comparator: Lamotrigine Brand | Experimental: Lamotrigine Generic
Number analyzed (Participants) | 4 | 4
ng*hr/ml | 79640 (11442) | 81653 (11991)

2. Primary Outcome: Cmax
Description: pharmacokinetic rate (ng/ml). Pharmacokinetic (PK) blood levels will be drawn at the schedule times: immediately prior to lamotrigine administration, then after drug administration at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, and 12.0 hr.
Time Frame: 0-12hr
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Active Comparator: Lamotrigine Brand | Experimental: Lamotrigine Generic
Number analyzed (Participants) | 4 | 4
ng/ml | 8836 (1245) | 9024 (1203)

ADVERSE EVENTS:
Arm/Group | Active Comparator: Lamotrigine Brand | Experimental: Lamotrigine Generic
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Comparator: Lamotrigine Brand (N=4) | Experimental: Lamotrigine Generic (N=4)
headache (Nervous system disorders) | 1 (2) | 2 (2)
dizziness (Nervous system disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This was a small study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes